CLINICAL TRIAL: NCT04910880
Title: Personal Protective Equipment Comfort and User Attitude During COVID-19 Pandemic: a Cross-Sectional Study Among Physical Therapy Students
Brief Title: Personal Protective Equipment Comfort and User Attitude During COVID-19
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 335561
Record Dates: First submitted 2021-05-29; First posted 2021-06-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Student; Physiotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
There are studies in the literature that evaluate the attitude, behavior and comfort level of students who do internships in different disciplines (medicine, pharmacy) towards the use of protective equipment. However, no study evaluating physiotherapy and rehabilitation students was found. Therefore, the present study aims to investigate the behaviors and attitudes regarding the use of personal protective equipment of physiotherapy and rehabilitation department students who are interning in the Covid-19 pandemic.

DETAILED DESCRIPTION:
A total of 250 participants, who are physiotherapy and rehabilitation intern students in Turkey, will be included in the present study. Data collection will be carried out using an online survey. The online survey link will be shared via social media accounts and via mail. The questionnaire created through Google forms will be delivered to the participants via the link. The link will be active in the data collection process. Before the participants start the questionnaire, they will be asked whether they were willing to participate. The socio-demographic characteristics (age, gender, weight, height) and health status (presence of chronic disease and drugs used) will be questioned. In addition, the information about the institution where the internship was held and the duration of the internship, internship hours, time spent at the internship will be collected. Personal Protective Equipment Comfort and User Attitude Evaluation Form will be used to evaluate participant's thoughts, attitudes and behaviors towards the use of personal equipment also physical complaints, comfort level due to personal protective equipment.

ELIGIBILITY:
Inclusion Criteria:

* The participants included in this study will be aged over 18 years, men or women, an intern student actively during Covid-19 pandemic and able to use computer and have an internet connection

Exclusion Criteria:

* Participants excluded from the study if they not able to understand and read Turkish as a language, do not use protective equipment with their own choice; do internship in a different discipline other than physiotherapy and rehabilitation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physical Therapy Students
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Evaluation Form | Baseline
  Demographic datas of the participants such as age, gender, height and weight will be recorded. At the same time, internship information and information about the use of personal protective equipment (mask, gloves, goggles, apron and overalls use) will be questioned.
The Attitude Inventory Regarding the Use of Personal Protective Equipment | Baseline
  There is no valid and reliable questionnaire evaluating behaviors and attitudes towards the use of personal protective equipment in the literature. Therefore, in our study, the attitudes and behaviors of the participants towards personal protective equipment will be evaluated using the questions developed in the article published by Çiriş et al. Required permissions have been obtained from the corresponding author of the article. "The Attitude Inventory Regarding the Use of Personal Protective Equipment" is composed of 5 likert scale type statements such as "1 - Strongly disagree," "2 - Disagree," "3 - Not sure," "4 - Agree," and "5 - Strongly agree." Answers to questions are between 1 and 5 points, so the total score varies between 5 and 100 points. As the score from each of the subgroups increases, the positive attitude toward the use of personal protective equipment increases.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No